CLINICAL TRIAL: NCT00875134
Title: Testing of the Apnea Prevention Device
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Mark H. Zornow, Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 10-06-54
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Respiratory Depression; Elective Surgery
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Verbal prompt, cutaneous stimulation (Experimental): Patient receives either or both a verbal stimulus or cutaneous stimulus
  Interventions: Other: Verbal prompt; Other: Skin Stimulus

INTERVENTIONS:
Other: Verbal prompt — Patient hears a voice recording
Other: Skin Stimulus — Patient receives either a skin stimulus

SUMMARY:
This study is designed to test the ability of a computer-based algorithm to detect and intervene in cases of narcotic-induced respiratory depression.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgical patients

Exclusion Criteria:

* Refusal to consent to study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2009-10 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Efficacy in treating respiratory depression | seconds after desaturation

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States